CLINICAL TRIAL: NCT01929668
Title: Comparison of 4L Polyethylene Glycol and 2L Polyethylene Glycol With Ascorbic Acid in Patients With Inactive Ulcerative Colitis; Randomized, Single Blind, Multicenter Study
Brief Title: Comparison of 4L Polyethylene Glycol and 2L Polyethylene Glycol With Ascorbic Acid in Inactive UC Patients
Acronym: 2SCANI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Eun Soo Kim, MD, PhD, Professor, Kyungpook National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 2013-07-036-002
Record Dates: First submitted 2013-08-23; First posted 2013-08-28 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Ulcerative Colitis
Keywords: ulcerative colitis; bowel preparation
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Polyethylene Glycols; Ascorbic Acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- polyethylene glycol (Active Comparator): 4L polyethylene glycol
  Interventions: Drug: polyethylene glycol
- polyethylene glycol with ascorbic acid (Experimental): 2L polyethylene glycol and ascorbic acid
  Interventions: Drug: polyethylene glycol; Drug: Ascorbic Acid

INTERVENTIONS:
Drug: polyethylene glycol
Drug: Ascorbic Acid
  Arms: polyethylene glycol with ascorbic acid

SUMMARY:
The purpose of this study is to compare preference of the patients, efficacy of preparation, and safety between 4 L polyethylene glycol and 2 L of polyethylene glycol with ascorbic acid in patients with inactive ulcerative colitis.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years old
* ulcerative colitis patients without symptoms for at least 1 year
* ulcerative colitis patients who undergo colonoscopy for surveillance

Exclusion Criteria:

* subjects who had abdominal surgery
* pregnant or breast feeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2013-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Number of patients who are willing to use the same preparation method for the next colonoscopy. | day 1

SECONDARY OUTCOMES:
Number of patients who have ulcerative colitis symptom aggravation within 30 days after bowel preparation, measured by simple clinical colitis activity index (SCCAI). | within 30 days after bowel preparation for colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Eun Soo Kim, MD, PhD, Principal Investigator — Keimyung University School of Medicine
Locations (1):
- Keimyung University Dongsan Medical Center, Daegu, South Korea